CLINICAL TRIAL: NCT06042374
Title: The Effects of Progressive Core Stabilization Training on Anaerobic Performance in Elite Athletes: A Randomized Controlled Trial.
Brief Title: Core Stabilization Training in Elite Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulsah Bargi (Other)
Responsible Party: Sponsor-Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Organization: Izmir Democracy University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Effect of core stabilization
Record Dates: First submitted 2023-08-30; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Athlete
Keywords: athlete; weightlifting; volleyball; racquet sports; core stability

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind study; the athletes were not informed about whether they were in the study group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The Progressive Core Stabilization Training was applied to study group as a group exercise with 5-10 athletes which was planned in the form of 3 days/week for a total of 9 weeks and 27 sessions.
  Interventions: Other: Progressive Core Stabilization Training
- Control group (Sham Comparator): The athletes included in the CG performed only Standard Core Strengthening Exercises.
  Interventions: Other: Standard Core Strengthening Exercises

INTERVENTIONS:
Other: Progressive Core Stabilization Training — The Progressive Core Stabilization Training was applied to study group as a group exercise with 5-10 athletes which was planned in the form of 3 days/week for a total of 9 weeks and 27 sessions. A session consisted of warm-up, core stabilization (30-40 min.), and cool-down exercises. During the training period, exercise volume, degree of difficulty, additional weight, and level of instability (contralateral limb movements and reduction of the support surface, etc.) for each exercise were incrementally increased in four steps.
  Arms: Study group
Other: Standard Core Strengthening Exercises — The athletes included in the CG performed only Standard Core Strengthening Exercises which is the first phase of the Progressive Core Stabilization Training on fixed surfaces (i.e. without pads and balls, with a flat floor and a bench) for 3 days/week and totally 9-week.
  Arms: Control group

SUMMARY:
The studies in the literature have not sufficiently investigated the effects of core stabilization training on anaerobic performance. Therefore, this study was planned to comparatively investigate effects of progressive core stabilization training applied to elite athletes on anaerobic capacity, anaerobic performance, and fatigue.

DETAILED DESCRIPTION:
In taekwondo, weightlifting, badminton, and volleyball sports branches, strong relationships between sports performance, anaerobic strength and fatigue parameters have been also shown. It is clear of the necessity of developing anaerobic capacity using various exercises in these elite athletes. However, the studies conducted to date have not sufficiently investigated the effects of core stabilization training on anaerobic performance and fatigue with more objective methods and enough sample sizes. This study was planned to comparatively investigate effects of progressive core stabilization training applied to elite athletes on anaerobic capacity, anaerobic performance, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* being between 18-25 of age,
* actively keeping on a similar technical workout season program,
* volunteering to participate in the study,
* having at least five years of professional sports history and
* being an elite athlete in taekwondo, weightlifting, volleyball, or badminton branches

Exclusion Criteria:

* having had any pathological condition and/or surgical procedure of the column vertebral and extremities within the last three months,
* having had any serious orthopedic or systemic condition that could prevent doing and continuing exercises
* discontinuing exercise training for more than three sessions.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
anaerobic peak power | Baseline and after 9-week training
  The power will be evaluated using anaerobic endurance test (a 30-second Wingate Anaerobic Power Test) applied on a bicycle ergometer.
anaerobic mean power | Baseline and after 9-week training
  The power will be evaluated using anaerobic endurance test (a 30-second Wingate Anaerobic Power Test) applied on a bicycle ergometer.

SECONDARY OUTCOMES:
squat jump power | Baseline and after 9-week training
  It will be evaluated the squat jump test.
active jump power | Baseline and after 9-week training
  It will be evaluated the active jump test.
fatigue index | Baseline and after 9-week training
  The percent of fatigue will be evaluated using anaerobic endurance test (a 30-second Wingate Anaerobic Power Test) applied on a bicycle ergometer.
anaerobic power from 0 to 5 seconds | Baseline and after 9-week training
  The power will be evaluated using anaerobic endurance test (a 30-second Wingate Anaerobic Power Test) applied on a bicycle ergometer.
anaerobic capacity from 0 to 30 seconds | Baseline and after 9-week training
  The power will be evaluated using anaerobic endurance test (a 30-second Wingate Anaerobic Power Test) applied on a bicycle ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BAŞANDAÇ, PhD., Principal Investigator — Mok Academy, Istanbul; GÜLŞAH BARĞI, Assoc. Dr., Principal Investigator — Izmir Democracy University; VOLGA BAYRAKCI TUNAY, Prof. Dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang CY, Thurston TS, Cho EH, Cho JY, Koo JH. Non-combative taekwondo evokes highly anaerobic physiological responses in elite-level athletes: potential evidence for a new training modality. J Sports Med Phys Fitness. 2019 Sep;59(9):1450-1457. doi: 10.23736/S0022-4707.18.09365-9. Epub 2018 Dec 13. PMID 30543275
- [Background] Lee B, McGill S. The effect of core training on distal limb performance during ballistic strike manoeuvres. J Sports Sci. 2017 Sep;35(18):1-13. doi: 10.1080/02640414.2016.1236207. Epub 2016 Oct 3. PMID 27690749
- [Derived] Basandac G, Bargi G, Bayrakci Tunay V. Effectiveness of progressive core stabilization training on anaerobic performance in elite athletes: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Aug 26;17(1):248. doi: 10.1186/s13102-025-01283-3. PMID 40859380